CLINICAL TRIAL: NCT06170463
Title: Combined Insulin Sensitizers as Double-Weapon to Detonate PCOS-induced Vicious Circle
Brief Title: Insulin Sensitizers Role in Control of PCOS Vicious Cycle.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Elnagar, Assistant professor of gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#11195-21/6-2023
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Met Group (Active Comparator)
  Interventions: Drug: Metformin Hydrochloride
- MI Group (Active Comparator)
  Interventions: Drug: MI/DCI combination in 40:1 ratio
- MM Group (Active Comparator)
  Interventions: Drug: Combination of Metformin hydrochloride and MI/DCI

INTERVENTIONS:
Drug: Metformin Hydrochloride — Met Group Received metformin hydrochloride 500 mg tab 3 times Daily
  Arms: Met Group
Drug: MI/DCI combination in 40:1 ratio — MI-group received MI/DCI combination in 40:1 ratio twice daily
  Arms: MI Group
Drug: Combination of Metformin hydrochloride and MI/DCI — MM Group Received both Met and MI Groups Treatment
  Arms: MM Group

SUMMARY:
PCOS is a common and complex disease affecting women of reproductive age. It is characterized by its complex pathological symptoms and mechanisms resulting in endocrine and metabolic dysfunction. PCOS is highly associated with various metabolic and endocrinal disorders. Metformin is mainly used for its glucose-lowering effects for treatment and prevention of type-2 diabetes mellitus (DM), gestational DM, and PCOS. Myo-inositol (MI) protects against MAFLD through reduction of hepatic accumulation of triglycerides.

ELIGIBILITY:
Inclusion Criteria:

* Age;
* Residence;
* level of education & type of work;
* Marital and fertility statuses, and if infertility was the main complaint;
* Presence of risk factors as sedentary lifestyle;
* Emotional stress and family history of PCOS;
* Obesity-related medical disorders especially DM or MAFLD;
* History of previous treatment for PCOS and its outcomes;
* Menstrual pattern such as infrequent menstrual periods.

Exclusion Criteria:

* Women had other manifestations of metabolic syndrome:
* Cardiac manifestations of PCOS;
* Maintained on other therapies or prepared for /received laparoscopic intervention for PCOS;
* Receiving scheduled exercise, lipid-lowering therapies, or maintained on diabetogenic drugs for any other indications;
* Had morbid obesity with body mass index (BMI) >35 kg/m2;
* Causes other than PCOS for infertility, manifest DM, hepatic or pancreatic diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Improvement of mensural pattern | 6 months
  The Evaluation of the success rate of the applied regimens to gain mensural regular pattern in PCOS Women

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Ash Sharqia Governorate, Egypt